CLINICAL TRIAL: NCT05237674
Title: MOVEOUT: a Cluster RCT of the Efficacy, Mechanisms, and Mediation of an Education Outside the Classroom Intervention on Adolescents' Physical Activity.
Brief Title: MOVEOUT: A Cluster RCT Investigating Education Outside the Classroom
Acronym: MOVEOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Center for Clinical Research and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2124712
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Psychological; Motivation; School Burnout
Keywords: School; Physical activity; Outdoor; Motivation; Education; Pedagogy; Wellbeing; Health Promotion
MeSH Terms: conditions — Sedentary Behavior; Burnout, Psychological; Motor Activity

STUDY DESIGN:
Intervention Model Description: Fifteen of thirty municipal primary and lower secondary schools with one or more classes in grade 4-10 will be randomly assigned to the TEACHOUT intervention. Classes within the other 15 schools will act as controls and continue their teaching as usual. Teachers of the participating classes in the waitlisted control schools will be offered the intervention once the trial is finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (Experimental): School children exposed to 1-2 weekly sessions, a total of at least five hours pr week, of education outside the classroom.
  Interventions: Behavioral: The TEACHOUT intervention
- Waiting control schools (No Intervention): The waiting control schools will receive the two-day training course on EOtC one year later immediately after post measurements are conducted.

INTERVENTIONS:
Behavioral: The TEACHOUT intervention — The core component of the Intervention is a two-day training course on EOtC given to elementary school teachers followed by the teachers committing to apply EOtC for at least five hours a week, delivered in 1-2 weekly sessions for one school year (in this study, August 2022 to June 2023).
  In the training course knowledge and understanding of the practice and theory of EOtC is facilitated in presentations and talks supplemented by illustrative examples in workshops and plenum discussions on local implementation. The 1-2 weekly EOtC sessions during the school year 2022-2023 may be delivered by one or more teachers simultaneously in various school subjects, at various places outside the school buildings.
  Arms: Intervention schools

SUMMARY:
The purpose of this study is to investigate the efficacy of an education outside the classroom (EOtC) intervention on adolescents' physical activity, school motivation, academic achievement, and wellbeing. The study will also investigate which pedagogical and didactical elements of EOtC are important to achieve more physical activity, school motivation, and wellbeing.

DETAILED DESCRIPTION:
Globally, many children and adolescents are insufficiently physically active which increases the prevalence of non-communicable diseases and poor mental health over the lifecourse. Schools are an important setting to promote physical activity (PA) as children and adolescents spend a large proportion of their waking hours in this setting. The MOVEOUT study aims to increase school-based PA and wellbeing trough implementing regular practice of education outside the classroom (EOtC) during school hours. In EOtC, teachers relocate teaching and learning activities to places and settings outside the school building, e.g., urban and green space, societal institutions, and private companies, in agreement with curricular aims, content and obligations. The aim of EOtC is to promote pupils' learning and wellbeing through practical activities and the use of body and senses in authentic situations. Cross-sectional studies suggest that practice of EOtC is positively associated with more moderate-to-vigorous PA for boys, and more and light-intensity PA for girls. Quasi-experimental studies further demonstrate a positive effect of regular practice of EOtC on school motivation and wellbeing, without compromising academic performance. However, no studies have investigated the effect of EOtC on PA, school motivation, or wellbeing in a randomised controlled design. Furthermore, the specific pedagogical and didactical elements in EOtC sessions that promote PA, school motivation, and wellbeing have not been researched. Therefore, the aim of MOVEOUT is to study the effect on adolescents' PA, school motivation, and wellbeing and the mechanisms of EOtC that might promote PA, school motivation, and wellbeing in a randomised controlled design.

Compared to previous studies, the MOVEOUT study provides a methodologically improved and more robust evaluation. This study investigates the efficacy, mechanisms, and mediating effects of an EOtC intervention, The TEACHOUT Intervention[1], in a cluster randomised waitlist controlled trial with 15 intervention schools and 15 control schools. Schools will be required to have one or more classes grade 4-10 (pupils aged 10-16). The study will investigate which pedagogical and didactical elements of EOtC that are important to achieve more PA, school motivation, and wellbeing for 1) all adolescents, 2) adolescents at risk of becoming overweight, and 3) boys and girls separately. MOVEOUT will provide solid evidence of the effect of EOtC and supplement theory on EOtC pedagogy and didactics, which is needed in practice and policy to inform the already ongoing scale-up of EOtC, for instance in Northern European countries. The study is conducted in partnership between the applying institutions and the participating schools through all phases.

ELIGIBILITY:
Inclusion Criteria

* Non-special need municipal primary and lower secondary school classes grade 4-10.
* Classes not involved in other school development or research projects.
* Participants for whom parents or legal guardians have provided written informed consent.
* Outcome data at baseline (for PA at least one time point; either winter or spring)

Exclusion Criteria

* Classes not able to comply with the following will be excluded from per-protocol analysis, but will be included in the intention-to-treat analysis: intervention group classes should have a school-year average of >150 min of weekly EOtC and the control group classes should have a school-year average of <=150 min of weekly EOtC.
* Pupils with significant health problems as judged by the investigators based on parents or legal guardians report of child health status will be excluded from the analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 1 school year
  Pupils' total daily time spent being sedentary, light, moderate and vigorous physically active and their daily time involved in running, walking, standing, sitting and lying will be measured with Axivity® AX3 accelerometers.
  All acceleration data will be processed in Matlab (Version 9.9.0 R2020b, Mathworks Inc., Natick, Massachusetts, US) which includes resampling, generating ActiGraph counts2, identification of non-wear, and summarising the subjects' time spent in different intensity domains. Non-wear periods will be identified from both acceleration and temperature data. PA will be measured two times (winter and spring) before the intervention (baseline) and the same time two times towards the end of the intervention (endline) to account for the context dependency of PA to seasonal conditions. The effect of the TEACHOUT intervention on PA intensities and behaviours will be investigated across two timeframes, i.e., during school hours and full days.
School motivation | 1 school year
  School motivation will be measured using the Academic Self-Regulation Questionnaire (called SRQ-A). The SRQ-A is a domain-specific self-report questionnaire developed for measuring the level of autonomy relative to doing different types of schoolwork among pupils in late primary and lower-secondary school.
Wellbeing | 1 school year
  Wellbeing will be measured using two different scales: KIDSCREEN-27 and the pro-social behaviour scales of Strengths and Difficulties Questionnaire (SDQ). KIDSCREEN-27 measures the subjective health and wellbeing or health-related quality of life of children and adolescents aged 8-18. The pro-social behaviour scale of the SDQ measures social skills and competences of adolescents. Data on school absence will be collected as an objective indicator of wellbeing.
Reading competence | 1 school year
  Reading competence will be measured with the validated age-adapted sentence reading test (Danish 'Sætningslæseprøve') by Hogrefe.
Mathematics skills | 1 school year
  Math skills will be measured with the validated age-adapted mathematical basic test (MG test in Danish) by Hogrefe.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Nielsen, PhD, Principal Investigator — University of Copenhagen; Mads Bølling, PhD, Study Director — Steno Diabetes Center Copenhagen; Peter Elsborg, PhD, Study Director — Center for Clinical Research and Prevention; Charlotte D Klinker, PhD, Study Chair — Steno Diabetes Center Copenhagen; Peter Bentsen, PhD, Study Chair — Center for Clinical Research and Prevention; Lærke M Grønfeldt, Msc, Study Director — Center for Clinical Research and Prevention
Locations (3):
- Denmark (3):
  - Center for Clinical Research and Prevention, Frederiksberg, Copenhagen
  - University of Copenhagen, Copenhagen
  - Steno Diabetes Center Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant-level data can be made available upon reasonable request to the PI such as e.g. verification of the research results. To comply with the European General Data Protection Regulation, and to accommodate article 10 of the Danish Act on Data Protection anonymised participant-level data will be made available on the Open Science Framework five years after the main publication of this study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anonymised participant-level data will be made available on the Open Science Framework five years after the main publication of this study.
  Statistical plan, study protocol and analytical code will be made available in the osf folder upon acceptance of first preregistered manuscript.
Access Criteria: Data can be made available upon reasonable request to the PI such as e.g. verification of the research results.
URL: https://osf.io/89pmf/?view_only=298a0d461e594bc3b2d73ace8d107882

REFERENCES:
- [Derived] Bolling M, Mygind L, Elsborg P, Melby PS, Barfod KS, Brond JC, Klinker CD, Nielsen G, Bentsen P. Efficacy and mechanisms of an education outside the classroom intervention on pupils' health and education: the MOVEOUT study protocol. BMC Public Health. 2023 Sep 19;23(1):1825. doi: 10.1186/s12889-023-16618-3. PMID 37726771